CLINICAL TRIAL: NCT04373200
Title: Human Ab Response & immunoMONItoring of COVID-19 Patients
Acronym: HARMONICOV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 35RC20_9795_HARMONICOV; 2020-A01100-39 (Other: ANSM (N°ID-RCB))
Record Dates: First submitted 2020-04-22; First posted 2020-05-04 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: SARS-CoV-2 Coronavirus; Acute Respiratory Distress Syndrome
Keywords: COVID-19; SARS-CoV-2 coronavirus; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19

STUDY DESIGN:
Intervention Model Description: Comparative study with 3 cohorts of 25 adult patients:
  * Cohort A: 25 COVID-19 associated ARDS
  * Cohort B: 25 COVID-19 without ARDS
  * Cohort C: 25 ARDS from other causes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- COVID-19 patients with associated ARDS (Experimental)
  Interventions: Biological: Blood samples collection; Other: Saliva collection
- COVID-19 patients without associated ARDS (Active Comparator)
  Interventions: Biological: Blood samples collection; Other: Saliva collection
- Patients with ARDS from other causes (Active Comparator)
  Interventions: Biological: Blood samples collection

INTERVENTIONS:
Biological: Blood samples collection — Blood sample collection at Day 1, day 7, day 14 for all patients. At month 4 for 25 survivors COVID-19 patients
Other: Saliva collection — Saliva collection at Month 4 for 25 survivors COVID-19 patients
  Arms: COVID-19 patients with associated ARDS; COVID-19 patients without associated ARDS

SUMMARY:
Prospective, mono centric study on COVID-19 patients with or without acute respiratory distress syndrome (ARDS) to analyse the dynamics of the immune response and to search for biomarkers of evolution

DETAILED DESCRIPTION:
Assessed by World Health Organisation as a pandemic on March 11, COVID-19 is caused by the SARS-CoV-2 coronavirus. The spectrum of its clinical manifestations is strikingly broad and extends from mild disease (resembling an ordinary bout of flu or even asymptomatic) to pneumonia. The latter cases convey a high risk of evolution towards acute respiratory distress syndrome (ARDS), eventually fatal when worsening with cytokine storm and multiple organ failure or with superinfection and sepsis. In the absence of overt variations of the virus itself, its interactions with the host immune system are likely crucial. Clinical features of patients with severe forms of COVID-19 were reported, but immunological description of biomarkers for exacerbation and mortality vs recovery remains superficial. Globally decreased white blood cells, notably T-cells, suggest that CoV-2 might trigger or exploit an immune defect. This could correspond to gaps in immune cell subpopulations, kinetics of activation or repertoires. Immune failure would then be responsible for exacerbations and a poor outcome in intensive care unit (ICU) patients. The objective of the study is to characterize the kinetics of the immune response and of immune dysregulation in ARDS patients. In addition to studying severe ARDS patients, an inverse image of immune repertoires should appear in healed up patients, after they have reached an undetectable viral load and acquired protective antibodies (Abs). Humoral immunity mediated by specific anti-viral Abs was a key factor for recovery from SARS-CoV-1 infection, and this is also expected for CoV-2, making the Ig repertoire also of special interest for its inclusion of anti-viral neutralizing Abs (nAbs).

Altogether, there is thus an urgent need for high-resolution characterization of the anti-CoV-2 immune response, correlating the dynamics of immune activation, cytokine production and immune repertoires with clinical evolution. In addition to providing biomarkers for prognosis evaluation and for monitoring innovative treatments this will also participate to the urgent quest of as many possible monoclonal antibodies (mAb) candidates for immunotherapy

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years old
* Patients COVID-19 :

  * hospitalized for less than 48 hours in intensive care unit (ICU) with ARDS (PaO2/Fi02 < 200) or
  * hospitalized with respiratory syndrome without need of invasive mechanical ventilation
* Patients hospitalized for less than 48 hours in intensive care unit (ICU) with ARDS (PaO2/Fi02 < 200) from other causes
* Patients who have given their consent or included in an emergency situation
* Patients affiliated to medical care insurance

Exclusion Criteria:

* Pregnant women
* Preexisting immune disorders (HIV-infection, malignancy, graft, treatment with immunosuppressive agents)
* Patients legally protected (under judicial protection, guardianship), persons deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-03-09 (Actual)

PRIMARY OUTCOMES:
Number of increased immune population | Month 4
  Blood sample
Number of decreased immune population | Month 4
  Blood sample
Number of statically different phenotypes compared to control patients | Month 4
  Blood sample

SECONDARY OUTCOMES:
Gain or loss of functional phenotypic markers between D1 and D14 | Day 14
  Qualitative identification of immune subpopulations showing a significant variation compared to controls and quantification of this variation (at D1 and/or D14)
Gain or loss of functional phenotypic markers between between acute and mild infections | Day 14
  Qualitative identification of immune subpopulations showing a significant variation between acute and mild COVID-19 and quantification of this variation (at D1 and/or D14)
Gain or loss of functional phenotypic markers between D1 and month 4 | Month 4
  Qualitative identification of immune subpopulations showing a significant variation between acute stage and recovery (at 4 months) and quantification of this variation
Evaluation of V, D, J gene usage alterations in the immunoglobulin and T cell receptor (TCR) repertoires during ARDS linked to COVID-19 | Day 14
  Blood sample
Identification of the Ig classes and of V, D, J sequences of anti-CoV-2 antibodies | Month 4
  Blood sample
Characterization of a new set of human antibodies from patients who have recovered of COVID-19 | Month 4
  Blood sample

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Pascal V, Dupont M, de Rouault P, Rizzo D, Rossille D, Jeannet R, Daix T, Francois B, Genebrier S, Cornic M, Monneret G, Venet F, Ferrant J, Roussel M, Reizine F, Le Souhaitier M, Tadie JM, Tarte K, Feuillard J, Cogne M. Demultiplexing Ig repertoires by parallel mRNA/DNA sequencing shows major differential alterations in severe COVID-19. iScience. 2023 Mar 17;26(3):106260. doi: 10.1016/j.isci.2023.106260. Epub 2023 Feb 21. PMID 36845033
- [Result] Roussel M, Ferrant J, Reizine F, Le Gallou S, Dulong J, Carl S, Lesouhaitier M, Gregoire M, Bescher N, Verdy C, Latour M, Bezier I, Cornic M, Vinit A, Monvoisin C, Sawitzki B, Leonard S, Paul S, Feuillard J, Jeannet R, Daix T, Tiwari VK, Tadie JM, Cogne M, Tarte K. Comparative immune profiling of acute respiratory distress syndrome patients with or without SARS-CoV-2 infection. Cell Rep Med. 2021 Jun 15;2(6):100291. doi: 10.1016/j.xcrm.2021.100291. Epub 2021 May 6. PMID 33977279
- [Derived] Hamzeh-Cognasse H, Mansour A, Reizine F, Mismetti P, Gouin-Thibault I, Cognasse F. Platelet-derived sCD40L: specific inflammatory marker for early-stage severe acute respiratory syndrome coronavirus 2 infection. Virol J. 2021 Oct 29;18(1):211. doi: 10.1186/s12985-021-01680-3. PMID 34715884